CLINICAL TRIAL: NCT05588570
Title: Coaching Children With Anxiety and Autism Through Telehealth
Acronym: CAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Laura Arnstein Carpenter, Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00121415
Record Dates: First submitted 2022-06-13; First posted 2022-10-20 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Autism; Autism Spectrum Disorder; Anxiety
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAT (Experimental): Participants will receive behavioral treatment for anxiety.
  Interventions: Behavioral: CAT

INTERVENTIONS:
Behavioral: CAT — Treatment includes 12 sessions: 2 caregiver teach sessions, 4 caregiver coach sessions in the child-directed interaction (CDI) phase, and 6 caregiver coach sessions in the DADS (Describe situation, Approach situation, give Direct command for child to join situation, provide Selective attention based on child's performance) phase. Throughout the 12 sessions, caregivers are coached through exposures in which the child is given the opportunity to slowly encounter anxiety-provoking factors. In the first session, caregivers are provided psychoeducation on anxiety and parenting practices and taught PRIDE (praise, reflect, imitate, describe, enjoy) skills, which are aimed at increasing approach behaviors and decreasing avoidant behaviors. In the CDI phase, caregivers are coached live via Bluetooth headset through the PRIDE and active ignoring skills. In the last 5 sessions, caregivers are coached through the DADS protocol while working up the Fear Hierarchy with the child.

SUMMARY:
This study will examine a telehealth parenting intervention to reduce anxiety in 20 families of children between 4 and 8 years old with autism and anxiety. Caregivers and children complete 12 telehealth treatment sessions. Caregivers and children will complete pre tests, post tests, and 3 month followup assessments that include observations, heart rate monitoring, and caregiver ratings.

DETAILED DESCRIPTION:
This study will examine the feasibility and initial efficacy of a telehealth adaptation of a parenting intervention to reduce anxiety (Coaching Approach behavior Leading by Modeling; CALM) amongst 20 families of children between 4 and 8 years old with autism and anxiety. Our time limited telehealth-delivered adaptation of CALM is called CAT (Coaching Children with Anxiety and Autism through Telehealth). The study will utilize an open trial design with pre, post, and 3-month follow-up assessments including observational measures, physiological measures, and caregiver ratings.

ELIGIBILITY:
Inclusion Criteria:

* Child participants must:
* Be between 4:0-8:11 years old
* Have clinically significant caregiver-report symptoms of anxiety on the Parent-Rated Anxiety Scale for ASD (PRAS-ASD)
* Have a primary anxiety concern on the Anxiety Disorders Interview Schedule for Autism Spectrum and Developmental Disorders: Parent Version (ADIS/ASA)
* Have an ASD diagnosis made by a qualified diagnostician
* Have a cognitive level of 48 months on the Wechsler Preschool & Primary Scale of Intelligence-Fourth Edition (WPPSI-IV; ages 2:6-7:7) or the Wechsler Intelligence Scale for Children-Fifth Edition (WISC-V; ages 6:0-16:11)

Caregiver participants must:

* Have access to a computer, tablet, or phone with a camera and Wi-Fi access

Exclusion Criteria:

* Primary concern other than anxiety as measures on the ADIS/ASA

Ages: 48 Months to 107 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Child Anxiety Symptoms as assessed by PRAS-ASD | Pre to Post (~14 weeks)
  The Parent Rated Anxiety Scale for ASD (PRAS-ASD) is a 25-item measure. Parents score severity of various anxiety symptoms on a scale of 0-3. The PRAS-ASD yields a total raw score for severity of anxiety and a normed T-score with higher scores indicating higher anxiety severity. The cut-off for clinical significance is a raw score of 44.
Change in Child Anxiety Symptoms as assessed by PRAS-ASD | Pre to Follow-up (~26 weeks)
  The Parent Rated Anxiety Scale for ASD (PRAS-ASD) is a 25-item measure. Parents score severity of various anxiety symptoms on a scale of 0-3. The PRAS-ASD yields a total raw score for severity of anxiety and a normed T-score with higher scores indicating higher anxiety severity. The cut-off for clinical significance is a raw score of 44.
Change in Parent Accommodation as assessed by FAS-A | Pre to Post (~14 weeks)
  The Family Accommodation Scale-Anxiety (FAS-A) is a 9 item measure. Parents score the amount that they accommodate their child's anxiety on a 0-4 frequency scale. The FAS-A yields a total raw score for accommodations and a normed T-score with higher scores indicating more accommodations.
Change in Parent Accommodation as assessed by FAS-A | Pre to Follow-up (~26 weeks)
  The Family Accommodation Scale-Anxiety (FAS-A) is a 9 item measure. Parents score the amount that they accommodate their child's anxiety on a 0-4 frequency scale. The FAS-A yields a total raw score for accommodations and a normed T-score with higher scores indicating more accommodations.
Child Heart Rate | Pre to Post (~14 weeks)
  Change in heart rate during structured play interaction from pre to post
Parent Heart Rate | Pre to Post (~14 weeks)
  Change in heart rate during structured play interaction from pre to post
Child Respiratory Sinus Arrhythmia as assessed by Actiheart software | Pre to Post (~14 weeks)
  Change in respiratory sinus arrhythmia during structured play interaction from pre to post while participant is wearing Actiheart electrodes. After heart activity is collected, Actiheart software is used to analyze Respiratory Sinus Arrhythmia (RSA)
Parent Respiratory Sinus Arrhythmia as assessed by Actiheart software | Pre to Post (~14 weeks)
  Change in respiratory sinus arrhythmia during structured play interaction from pre to post while participant is wearing Actiheart electrodes. After heart activity is collected, Actiheart software is used to analyze Respiratory Sinus Arrhythmia (RSA)
Parent Anxiety Symptoms as assessed by GAD-7 | Pre to Post (~14 weeks)
  The Generalized Anxiety Disorder (GAD-7) is a 7-item screening tool to assess for adult anxiety. Parents score their anxiety symptoms on a 0-3 frequency scale. The GAD-7 yields a total raw score for level of anxiety and a normed T-score with higher scores indicating higher levels of anxiety. The cut-off for clinical significance is a raw score of 8.
Parent Anxiety Symptoms as assessed by GAD-7 | Pre to Follow-up (~26 weeks)
  The Generalized Anxiety Disorder (GAD-7) is a 7-item screening tool to assess for adult anxiety. Parents score their anxiety symptoms on a 0-3 frequency scale. The GAD-7 yields a total raw score for level of anxiety and a normed T-score with higher scores indicating higher levels of anxiety. The cut-off for clinical significance is a raw score of 8.
Change in Parenting Stress as assessed by Parenting Stress Index-Short Form (PSI-SF) | Pre to Post (~14 weeks)
  Parents will complete the PSI-SF, a 36-item measure yielding scores for a Total Stress scale. The PSI-SF is a widely used measure in ASD samples and has been used as an outcome measure in PCIT ASD studies. The PSI-SF yields a total raw score for stress level and a percentile score which describes parent stress relative to all parents assessed during the development and testing of the PSI. Scores above 80 are considered high stress scores.
Change in Parenting Stress as assessed by Parenting Stress Index-Short Form (PSI-SF) | Pre to Follow (~26 weeks)
  Parents will complete the PSI-SF, a 36-item measure yielding scores for a Total Stress scale. The PSI-SF is a widely used measure in ASD samples and has been used as an outcome measure in PCIT ASD studies. The PSI-SF yields a total raw score for stress level and a percentile score which describes parent stress relative to all parents assessed during the development and testing of the PSI. Scores above 80 are considered high stress scores.

SECONDARY OUTCOMES:
Caregiver Satisfaction with treatment as assessed by Therapy Attitude Inventory (TAI) | Pre to Post (~14 weeks)
  To assess treatment satisfaction, parents will complete the TAI, which is widely used in PCIT studies. Several questions will be added to the TAI to address parental satisfaction and openness regarding the telehealth delivery format for families in the Tele-PCIT condition. The TAI uses a Likert-type satisfaction scale and scores will be reported via descriptive statistics with 95% CIs within categories.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No